CLINICAL TRIAL: NCT05481086
Title: The Effects Pain Severity on Individuals With Fibromyalgia Syndrome
Brief Title: Pain Severity in Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Director, Kutahya Health Sciences University
Other Study IDs: Fibromyalgia pain insenty
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Fibromyalgia; Pain, Chronic
Keywords: fibromyalgia; pain; patient reported outcome measurement
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Individuals with fibromyalgia syndrome
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — There is no interventions in this study

SUMMARY:
Fibromyalgia Syndrome (FMS) is a complex syndrome that mainly includes the musculoskeletal system and is characterized by many symptoms such as chronic widespread pain, fatigue and sleep disorders, cognitive dysfunctions, regional pain syndrome, psychiatric disorders. The existence and importance of the multidimensional nature of chronic pain in FMS has been demonstrated. Factors such as pain intensity, persistence of pain, pain-related disability, and novelty of onset are all important characteristics of a chronic pain condition. Therefore, there was a need for a global measure of chronic pain severity that summarized different measures of pain and a graded classification of chronic pain was proposed. Patients with chronic pain such as FMS are known to have a greater negative impact than many chronic medical conditions. Chronic pain severity in FMS has been found to be associated with various conditions such as function and health status, and it has been shown that reduction in pain severity provides broadly beneficial results on these conditions. However; there are no studies in which chronic pain severity in FMS is classified by grading and investigating the relationship of different pain severity degrees with disease severity and other symptoms.

The aim of this study is to evaluate whether the severity of the disease, kinesiophobia, and concerns about pain differ in individuals with different pain severity by grading the severity of pain in individuals with fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* to be aged between 18-65,
* to be diagnosed with fibromyalgia syndrome according to the criteria of 2016 ACR
* to be volunteer to participate in the study.

Exclusion Criteria:

* Having cognitive impairment
* Illiterate people
* Diagnosed severe mental and psychological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who directly presented to the Physical Therapy Department of Kutahya Health Sciences University Hospital during the study period (between 15 August and 15 Nowember) with persistent and diffuse pain, will be screened for eligibility by an independent physician (M.A.L.)
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Chronic Pain Grading Scale-Revised (CPGS-R) | 5 minutes
  Pain severity and degree will be evaluated with the "Revised Graded Chronic Pain Scale (GCPS-R)". The "Graded Chronic Pain Scale" was created by Von Korff et al (1) to evaluate the severity of pain and disability related to pain in individuals with chronic pain. It has also been revised by the same authors (2). The Turkish validity and reliability study of the GCPS-R was performed by Özden et al (3).
Revised Fibromyalgia Impact Questionnaire | 10 minutes
  The Fibromyalgia Impact Questionnaire was developed by Burckhardt et al (4). The scale was revised by Bennett et al (5). The Turkish validity and reliability study of the FIQ-R was performed by Ediz et al (6). The structure of the FIQ-R's original questionnaire, based on function, overall effect, and severity of FM symptoms (disease severity) is the same as in the FIQ. However, questions assessing altered function, which were not part of the original FIQ, and questions measuring cognitive impairment, sensitivity, balance, and environmental sensitivity have been added to the FIQ-R. Also, some of the wording, missings, concepts and scoring problems in the original FIQ have been corrected in the FIQ-R. FIQ-R consists of 21 questions in total.
Tampa Kinesiophobia Scale | 10 minutes
  "Tampa Kinesiophobia Scale (TKS)" will be used to evaluate kinesiophobia. The Turkish version was created by Yılmaz et al (7). The scale consists of 17 questions developed to measure the fear of movement and/or re-injury.
UW-Concerns About Pain | 5 minutes
  Participants' pain concerns will be assessed with the "University of Washington Concerns About Pain (UWCAP)", which was recently developed as a pain self-efficacy measure based on modern scale development approaches. The scale was adapted to Turkish by Saraçoğlu et al (UWCAP-TR-6). "UWCAP-TR-6" consists of 6 questions.

SECONDARY OUTCOMES:
Short form-12 (SF-12) questionnaire | 5 minutes
  Turkish Short form-12 (SF-12) questionnaire, 12-item generic self-administered instrument that consists of eight subscales relating to various aspects of the QoL: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: İSMAİL SARAÇOĞLU, Ph.D., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University Evliya Celebi Hospital Physical Therapy and Rehabilitation Department, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No